CLINICAL TRIAL: NCT02874183
Title: Pharmacist Role in HF Patients Transition of Care: Randomized Clinical Trial (RCT)
Brief Title: Pharmacist Role in HF Patients Transition of Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborating site had difficulty with approval
Sponsor: Nova Southeastern University (Other)
Collaborators: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Fatimah M. Sherbeny, PharmD,MS., Ph.D. candidate at Nova Southeastern University - College of Pharmacy, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-052
Record Dates: First submitted 2016-08-02; First posted 2016-08-22 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; HF; CHF; RCT; Self-efficacy; Pharmacy; Pharmacist; Transition of Care; Readmission
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist intervention group (Experimental): The intervention group will receive:
  1. A phone call 48h-72h after discharge from the hospital to ensure that the patient filled their prescriptions and started taking their medication.
  2. A phone call five to seven days after discharge to reinforce the education using the "teach back technique"1. Patients will be asked about their medications, what are they for, how to use them, and what side effects to watch for, based on the education and information that was provided to them at discharge.
  Interventions: Behavioral: Pharmacist intervention
- usual care group (No Intervention): The control group will receive the usual standard care available at West Kendall Baptist Hospital.

INTERVENTIONS:
Behavioral: Pharmacist intervention — Pharmacist counseling and follow-up phone calls
  Arms: Pharmacist intervention group

SUMMARY:
To assess the effectiveness of pharmacist's provided education in HF patients, in improving patients' knowledge and self-efficacy, and to assess the impact of this intervention on the rate of hospital readmission and emergency visits at 30-days, 60-days and 90-days after discharge.

DETAILED DESCRIPTION:
"Transition of care" is one of the new disciplines that pharmacists have been involved-in within the healthcare system. It is a process where a patient's care is shifting from one setting to another. During this process, transitional care is designed to ensure continuity of patient care across different sites or across different levels of care within the same facility. For example, from Intensive Care Unit (ICU) to the ward, from hospital to home, or from hospital to rehab centers. Many stakeholders are involved in this process, and coordination between them is necessary to have successful one, in addition to logistical arrangements, and patient education. Otherwise, poor communication, inadequate patient education, and lack of access to healthcare services, will produce failure of having a smooth transition and could result in negative health outcomes including complications in the patient's disease status, emergency room visits or hospital readmissions. Not only that these negative health outcomes are affecting the patient, they are also negatively affecting the healthcare spending in the United States. For instance, inadequate care coordination and management of care transitions accounted for $25 to $45 billion in wasteful spending in 2011 through preventable adverse events and hospital readmissions. Therefore, cost containment and reducing the excessive spending in healthcare is an important aim of "transition of care", secondary to improving patient outcomes.

Pharmacist's role in Transition of care:

Pharmacists have the knowledge, training and expertise to play a major role in the transition of care process. They are involved in dispensing the patient's medications at the hospital, ensuring that the patient's medication chart is updated, identify any medication discrepancy, provide medication reconciliation, medication education, patient counseling at discharge and they could follow-up with the patients after discharge to check if they filled their prescription, what side effects are they having, and monitor their adherence to their treatment plan. These pharmacist's interventions have been applied, among other approaches, by hospitals to improve the quality of their services and minimize the rate of readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted HF patients at WKBH
* Patients with primary or secondary diagnosis of HF
* Discharged to Home
* 18 years old or older

Exclusion Criteria:

* ≥ 90 years old
* Patients with major comorbidities such as cancer, end-stage kidney disease, and liver failure
* Patients with memory problems such as dementia and Alzheimer's disease
* Patients discharged to places other than home
* Patients who are unable to understand or follow discharge instructions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change in knowledge | at baseline, 30 days, 60 days and 90 days after hospital discharge
  The investigators will measure patient's knowledge about heart failure using a 15 item questionnaire, at baseline (at recruitment) before they get the discharge counseling at West Kendall Baptist Hospital (WKBH), then the investigators will measure it again 30 days, 60 days, and 90 days after discharge to evaluate the change in the patient's knowledge and how much information did the patients retain after the discharge counseling.
change in self-efficacy using a 16 items scale | at baseline, 30 days, 60 days and 90 days after hospital discharge
  the investigators will measure patient's self-efficacy, using a 16 items scale, at baseline (at recruitment) before the patients get the discharge counseling at West Kendall Baptist Hospital (WKBH), then the investigators will measure it again 30 days, 60 days, and 90 days after discharge to evaluate the change in the patient's self-efficacy and ability to take care of themselves before and after they receive the discharge counseling and be educated about heart failure and how to manage it.

SECONDARY OUTCOMES:
hospital readmission rate | 30 days after hospital discharge
hospital readmission rate | 60 days after hospital discharge
hospital readmission rate | 90 days after hospital discharge
number of emergency visits | 30 days after hospital discharge
number of emergency visits | 60 days after hospital discharge
number of emergency visits | 90 days after hospital discharge

REFERENCES:
- [Background] Coleman EA. Falling through the cracks: challenges and opportunities for improving transitional care for persons with continuous complex care needs. J Am Geriatr Soc. 2003 Apr;51(4):549-55. doi: 10.1046/j.1532-5415.2003.51185.x. PMID 12657078
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Aminzadeh F, Dalziel WB. Older adults in the emergency department: a systematic review of patterns of use, adverse outcomes, and effectiveness of interventions. Ann Emerg Med. 2002 Mar;39(3):238-47. doi: 10.1067/mem.2002.121523. PMID 11867975
- [Background] Hawes EM, Maxwell WD, White SF, Mangun J, Lin FC. Impact of an outpatient pharmacist intervention on medication discrepancies and health care resource utilization in posthospitalization care transitions. J Prim Care Community Health. 2014 Jan 1;5(1):14-8. doi: 10.1177/2150131913502489. Epub 2013 Sep 17. PMID 24327590
- [Background] Bellone JM, Barner JC, Lopez DA. Postdischarge interventions by pharmacists and impact on hospital readmission rates. J Am Pharm Assoc (2003). 2012 May-Jun;52(3):358-62. doi: 10.1331/JAPhA.2012.10172. PMID 22618976
- [Background] Thomas R, Huntley AL, Mann M, Huws D, Elwyn G, Paranjothy S, Purdy S. Pharmacist-led interventions to reduce unplanned admissions for older people: a systematic review and meta-analysis of randomised controlled trials. Age Ageing. 2014 Mar;43(2):174-87. doi: 10.1093/ageing/aft169. Epub 2013 Nov 5. PMID 24196278